CLINICAL TRIAL: NCT05116150
Title: Effects of Combined Grape Seed Extract and L-citrulline Supplementation on Hemodynamic Responses in Young Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California Baptist University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 112-1819 EXP
Record Dates: First submitted 2021-10-19; First posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Dietary Supplementation
MeSH Terms: interventions — Grape Seed Extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Randomized double blind grape seed extract design (Active Comparator): Grape see extract
  Interventions: Dietary Supplement: Grape seed extract; Dietary Supplement: Placebo
- Randomized double blind placebo design (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Grape seed extract; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Grape seed extract — Effects of 7 days of combined GSE with L-citrulline supplementation on hemodynamic responses at rest and during cycling exercise.
Dietary Supplement: Placebo — Effects of 7 days of placebo supplementation on hemodynamic responses at rest and during cycling exercise.

SUMMARY:
This study was to examine the additive benefits with combined grape seed extract (GSE) and L-citrulline supplementation on hemodynamic responses to dynamic exercise, 11 young, healthy males were recruited for this study.

DETAILED DESCRIPTION:
The investigators aimed the additive effects of combined grape seed extract (GSE) and L-citrulline supplementation on hemodynamic responses to dynamic exercise, 11 young, healthy males were recruited for this study. Effects of 7 days of combined GSE with L-citrulline supplementation on systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial blood pressure (MAP), cardiac output (CO), total vascular conductance (TVC), and oxygen consumption (O2) were examined at rest and during cycling exercise.

ELIGIBILITY:
Inclusion Criteria:

* healthy males

Exclusion Criteria:

* cardiovascular and/or pulmonary disease, musculoskeletal disorders, or medications that prevent the safe completion of the exercise protocol

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure (mmHg) | 7 days
  by sphygmomanometer
Diastolic blood pressure (mmHg) | 7 days
  by sphygmomanometer
Mean arterial pressure (mmHg) | 7 days
  calculated (MAP = (SBP-DBP)/3 + DBP
Heart rate (bpm) | 7 days
  measured using Physio Flow (non-invasive device)
Stroke volume (ml) | 7 days
  measured using Physio Flow (non-invasive device)
Cardiac output (l/min) | 7 days
  calculated: HR (bpm) x SV (ml)
Total vascular conductance (ml/min/mmHg) | 7 days
  calculated: CO (ml/min) / MAP (mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Kyung Kim, Ph.D, Principal Investigator — California Baptist University
Locations (1):
- California Baptist University, Riverside, California, United States

IPD SHARING:
Plan to Share IPD: Undecided